CLINICAL TRIAL: NCT06206408
Title: A Phase 3, Randomized, Placebo-controlled, Double-blind Study to Assess the Efficacy and Safety of Fezolinetant in Japanese Women Experiencing Vasomotor Symptoms (Hot Flashes) Associated With Menopause
Brief Title: A Study to Confirm if Fezolinetant Helps Reduce Hot Flashes in Japanese Women Going Through Menopause
Acronym: Starlight 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2693-CL-0310; jRCT2031230571 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hot Flashes
Keywords: menopause;; ESN364;; vasomotor symptoms;; fezolinetant;; VEOZAH™
MeSH Terms: conditions — Hot Flashes | interventions — fezolinetant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fezolinetant low dose (Experimental): Participants will receive low dose of fezolinetant and placebo once daily for 12 weeks.
  Interventions: Drug: Fezolinetant; Drug: Placebo
- Fezolinetant high dose (Experimental): Participants will receive high dose of fezolinetant and placebo once daily for 12 weeks.
  Interventions: Drug: Fezolinetant; Drug: Placebo
- Placebo (Placebo Comparator): Participants will receive matching placebo once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fezolinetant — oral
  Other Names: ESN364;; VEOZAH™
  Arms: Fezolinetant high dose; Fezolinetant low dose
Drug: Placebo — oral

SUMMARY:
Hot flashes are the most common reason women going through menopause seek medical attention. Hormone replacement therapy, or HRT, is most often prescribed to treat hot flashes. However, HRT can't be used by all women or for as long as may be needed.

Researchers want to find other ways to treat hot flashes. Fezolinetant is a medicine to treat hot flashes in women going through menopause. Fezolinetant is an approved medicine in the US. Further studies are needed before it is available in other regions such as Asia.

This study will confirm if fezolintant helps reduce the number of hot flashes in Japanese women going through menopause.

Women that want to take part in the study will be given an electronic handheld device with an app to track their hot flashes. Some women may be able to use the app on their own smartphone. Before the women are assigned a treatment, they will record information about their hot flashes.

Women will either take a lower or higher dose of fezolinetant, or a placebo. This is decided by chance alone. The placebo looks like fezolinetant but will not have any medicine in it.

The women will take 2 tablets of the study medicine (lower or higher dose of fezolinetant, or the placebo) once a day for up to 12 weeks. They will either take 1 tablet of fezolinetant (higher or lower dose) and 1 placebo tablet, or they will take 2 placebo tablets. The women will continue to record information about their hot flashes on the electronic device or their smartphone.

During the study, the women will visit the study clinic a few times. At each visit they will be asked if they had any medical problems and will use an electronic device at the clinic to answer questions about how the hot flashes affect their daily life. Other checks will include a medical examination, vital signs (temperature, blood pressure and pulse). Some blood and urine samples will be taken for laboratory tests. At some visits, the women will also have an ECG to check their heart rhythm. Women who have a womb (uterus) will also have a test called a transvaginal ultrasound. A probe is gently placed inside the vagina. Sound waves will create a picture of the organs in the pelvis. This will allow the study doctor to look more closely at the uterus and surrounding organs.

The last clinic visit will be 3 weeks after the women take their final tablets of the study medicine (1 tablet of lower or higher dose of fezolinetant and 1 placebo tablet, or 2 placebo tablets).

ELIGIBILITY:
Inclusion Criteria:

* Participant confirmed as menopausal per one of the following criteria at the screening visit (visit 1):

  * Spontaneous amenorrhea for >/=12 consecutive months;
  * Spontaneous amenorrhea for >/=6 months with biochemical criteria of menopause (follicle-stimulating hormone (FSH) > 40 IU/L);
  * Having had bilateral oophorectomy >/=6 weeks prior to the screening visit (visit 1) (with or without hysterectomy); or
  * Having had hysterectomy without bilateral oophorectomy with the biochemical criteria of menopause (FSH > 40 IU/L).
* Participant must be seeking treatment or relief for vasomotor symptoms (VMS) associated with menopause and meet some set criteria related to hot flash(es) (HFs) (VMS) prior to randomization.
* Participant agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Participant has a history of an undiagnosed uterine bleeding within the 6 months prior to the screening visit (visit 1).
* Participant has a current malignant tumor or history (except for a participant who has not received treatment for malignant tumors for at least 5 years before informed consent acquisition and was not considered to have recurrence) of a malignant tumor except for non-metastatic basal cell carcinoma of the skin.
* Participant has a medical condition or chronic disease (including history of neurological [including cognitive], hepatic, renal, cardiovascular, gastrointestinal, pulmonary [e.g., moderate asthma], endocrine, or gynecological disease) that could confound interpretation of the study outcome.
* Participant uses a prohibited therapy (hormone therapy, hormone replacement therapy (HRT), hormonal contraceptive, any treatment for menopausal symptoms [prescription medications, over-the-counter, or herbal/Kampo medicines] or strong or moderate cytochrome P450 1A2 (CYP1A2) inhibitors) and is not willing to wash out or discontinue use of such drugs from screening visit (visit 1) through the follow-up visit (visit 6) or it is not medically appropriate to discontinue such drugs for the duration of the study.
* Participant has been randomized/registered in a clinical study with fezolinetant previously or had previous exposure to marketed fezolinetant elsewhere.
* Participant has a present or previous history of participation in this study.
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening (visit 1).
* Participant has an unacceptable result from the transvaginal ultrasound (TVU) assessment at screening (i.e., full length of endometrial cavity cannot be visualized or presence of clinically significant abnormal findings).
* Participant has documentation of a clinically significant abnormal Papanicolaou (Pap) test (or equivalent cervical cytology) within the 12 months prior to the screening visit (visit 1) or at screening.
* Participant has active liver disease, jaundice, or elevated liver aminotransferases (alanine aminotransferase (ALT) or aspartate aminotransferase (AST)), elevated total bilirubin (TBL) or direct bilirubin (DBL), elevated international normalized ratio (INR), or elevated alkaline phosphatase (ALP) at screening. A participant with mildly elevated ALT or AST up to < 1.5 × upper limit of normal (ULN) can be enrolled if TBL and DBL are normal. Participant with mildly elevated ALP (up to < 1.5 × ULN) can be enrolled if cholestatic liver disease is excluded and no cause other than fatty liver is diagnosed. Participant with Gilbert's syndrome with elevated TBL may be enrolled as long as DBL, hemoglobin and reticulocytes are normal.
* Participant has creatinine > 1.5 × ULN or estimated glomerular filtration rate using the Modification of Diet in Renal Disease formula </=30 mL/min/1.73 m^2 at screening.
* Participant has positive hepatitis serology panel (i.e., positive hepatitis B surface (HBs) antigen and/or positive hepatitis C virus (HCV) antibody) at screening. If HCV antibody test result is equivocal, hepatitis C virus ribonucleic acid (HCV RNA) test at study site is allowed. Participant can be enrolled if that result is normal or not abnormal.
* Participant is not in good general health as determined on the basis of medical history and general physical examination performed at the screening; hematology parameters, biochemistry parameters, pulse rate, blood pressure, electrocardiogram (ECG) outside the reference range for the population studied, or is showing clinically relevant deviations.
* Participant has a history of suicide attempt or suicidal behavior within the 12 months prior to study enrollment or suicidal ideation within the 12 months prior to study enrollment (a response of "yes" to question 4 or 5 on the suicidal ideation portion of the Columbia Suicide Severity Rating Scale (C-SSRS)), or is at significant risk to commit suicide at day 1 (visit 2).
* Participant is unable or unwilling to complete the study procedures.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to fezolinetant or any components of the formulation used.
* Participant is the investigator or a member of the study site staff.
* Participant is an employee of Astellas, the study-related contract research organizations (CROs) or site management organization.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in the frequency of mild to severe vasomotor symptoms (VMS) | Baseline and Week 8
  Frequency of mild, moderate or severe VMS events will be calculated as the sum of mild, moderate or severe VMS events per day.

SECONDARY OUTCOMES:
Mean change from baseline in the frequency of mild to severe VMS | Baseline and up to Week 12
  Frequency of mild, moderate or severe VMS events will be calculated as the sum of mild, moderate or severe VMS events per day.
Mean change from baseline in the frequency of moderate to severe VMS | Baseline and up to Week 12
  Frequency of moderate or severe VMS events will be calculated as the sum of moderate or severe VMS events per day.
Mean percent reduction in the frequency of mild to severe VMS from baseline | Baseline and up to Week 12
  Frequency of mild, moderate or severe VMS events will be calculated as the sum of mild, moderate or severe VMS events per day. Mean percent reduction will be reported.
Mean percent reduction in the frequency of moderate to severe VMS from baseline | Baseline and up to Week 12
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate or severe VMS events per day. Mean percent reduction will be reported.
Percent reduction of >/= 50% in the frequency of mild to severe VMS from baseline | Baseline and up to Week 12
  Frequency of mild, moderate or severe VMS events will be calculated as the sum of mild, moderate or severe VMS events per day. Percent reduction of >/= 50% will be reported.
Percent reduction of >/= 75% in the frequency of mild to severe VMS from baseline | Baseline and up to Week 12
  Frequency of mild, moderate or severe VMS events will be calculated as the sum of mild, moderate or severe VMS events per day. Percent reduction of >/= 75% will be reported.
Percent reduction of 100% in the frequency of mild to severe VMS from baseline | Baseline and up to Week 12
  Frequency of mild, moderate or severe VMS events will be calculated as the sum of mild, moderate or severe VMS events per day. Percent reduction of 100% will be reported.
Percent reduction of >/= 50% in the frequency of moderate to severe VMS from baseline | Baseline and up to Week 12
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate or severe VMS events per day. Percent reduction of >/= 50% will be reported.
Percent reduction of >/= 75% in the frequency of moderate to severe VMS from baseline | Baseline and up to Week 12
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate or severe VMS events per day. Percent reduction of >/= 75% will be reported.
Percent reduction of 100% in the frequency of moderate to severe VMS from baseline | Baseline and up to Week 12
  Frequency of moderate and severe VMS events will be calculated as the sum of moderate or severe VMS events per day. Percent reduction of 100% will be reported.
Number of participants with Adverse Events (AEs) | Up to Week 15
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures.
Change from baseline in endometrial thickness | Baseline and up to Week 12
  Endometrial thickness is a measure of how thick the lining of the uterus is. Endometrial thickness will be measured by transvaginal ultrasound (TVU).
Number of participants with laboratory value abnormalities and/or AEs | Up to Week 15
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or AEs | Up to Week 15
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to Week 12
  Number of participants with potentially clinically significant ECG values.
Pharmacokinetics (PK) of fezolinetant in plasma: Concentration | Up to Week 12
  Concentration will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of metabolite ES259564 in plasma: Concentration | Up to Week 12
  Concentration will be recorded from the PK plasma samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Study Director — Astellas Pharma Inc
Locations (64):
- Japan (64):
  - Chita Kosei Hospital, Chita-gun, Aichi-ken
  - Konan Kosei Hospital, Kōnan, Aichi-ken
  - Daido Clinic, Nagoya, Aichi-ken
  - MEITETSU Hospital, Nagoya, Aichi-ken
  - Toyota Kosei Hospital, Toyota-shi, Aichi-ken
  - Chiba Aoba Municipal Hospital, Chiba, Chiba
  - Aiiku Ladies Clinic, Funabashi-shi, Chiba
  - Tsujinaka Hospital Kashiwanoha, Kashiwa-shi, Chiba
  - Juno Vesta Clinic hatta, Matsudo-shi, Chiba
  - Fukuoka Mirai Hospital, Fukuoka, Fukuoka
  - Mori Ladies Clinic, Fukuoka, Fukuoka
  - Nishiguchi Clinic Fujinka, Fukushima, Fukushima
  - National Hospital Organization Takasaki General Medical Center, Takasaki-shi, Gunma
  - Sato Hospital, Takasaki-shi, Gunma
  - Sadamori Ladies Clinic, Hiroshima, Hiroshima
  - Kotoni Ladies Clinic, Sapporo, Hokkaido
  - M's Ladies Clinic, Sapporo, Hokkaido
  - Miyanomori Ladies' Clinic, Sapporo, Hokkaido
  - Social Medical Corporation Caress Sapporo Caress Memorial Hospital, Sapporo, Hokkaido
  - Kosumo Clinic, Kako-gun, Hyōgo
  - Mari Women'S Clinic, Nisinomiya-shi, Hyōgo
  - JA Toride Medical Center, Toride, Ibaraki
  - Tsukuba Urocare Clinic, Tsukuba, Ibaraki
  - National Hospital Organization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Asahi Clinic, Takamatsu, Kagawa-ken
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Kawasakieki Fumi Ladies Clinic, Kawasaki-shi, Kanagawa
  - Koukan Clinic, Kawasaki-shi, Kanagawa
  - Shinkawasaki Kobiki Womens Clinic, Kawasaki-shi, Kanagawa
  - Motomachi Ladies Clinic, Yokohama, Kanagawa
  - Women's Clinic LUNA Yokohama Motomachi, Yokohama, Kanagawa
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - Chieko Yukika Lady's Clinic, Sendai, Miyagi
  - Social Medical Care Corporation Hosei-kai Marunouchi Hospital, Matsumoto-shi, Nagano
  - National Hospital Organization Beppu Medical Center, Beppu-shi, Oita Prefecture
  - Miyabi Uro-Gyne Clinic, Okayama, Okayama-ken
  - National Hospital Organization Osaka Minami Medical Center, Kawachinagano-shi, Osaka
  - Chayamachi Ladies Clinic, Osaka, Osaka
  - Chiharu Clinic, Osaka, Osaka
  - GyNet Medical Corporation Minamimorimachi Ladies' Clinic, Osaka, Osaka
  - Kitahorie Kanade Ladies Clinic, Osaka, Osaka
  - Komorebi Ladies Clinic Osaka Honmachi, Osaka, Osaka
  - Ninomiya Ladies Clinic, Osaka, Osaka
  - Rikako Ladies Clinic, Osaka, Osaka
  - Tennoji Chihiro Women's Clinic, Osaka, Osaka
  - Shimizu Ladies Clinic, Sakai-shi, Osaka
  - jMOG Medical Corporation Tanabe Ladies' Clinic, Takatsuki-shi, Osaka
  - OHARA Clinic, Saitama, Saitama
  - Maruyama Memorial General Hospital, Saitama-shi, Saitama
  - Omi Medical Center, Social Medical Corporation Seikoukai, Kusatsu-shi, Shiga
  - Omihachiman Community Medical Center, Ōmihachiman, Shiga
  - Sei Women's Clinic, Bunkyo-ku, Tokyo
  - Marunouchi no Mori Ladies Clinic, Chiyoda-ku, Tokyo
  - Medical Corporation Asbo Tokyo Asbo Clinic, Chuo-ku, Tokyo
  - Medical Corp. SEIKOUKAI New Medical Research System Clinic, Hachioji-shi, Tokyo
  - Machida Municipal Hospital, Machida-shi, Tokyo
  - Toranomon Womens Clinic, Minato-ku, Tokyo
  - Kichijyoji Ladies Clinic, Musashino-shi, Tokyo
  - Shimamura Memorial Hospital, Nerima-ku, Tokyo
  - Yukawa Women'S Clinic, Nishi-Tokyo-shi, Tokyo
  - Shimodaira Ladies Clinic, Suginami-ku, Tokyo
  - Medical Corporation Associa Tamacenter Ladies Clinic, Tama-Shi, Tokyo
  - Japan Community Health care Organization Tokuyama Central Hospital, Shunan-shi, Yamaguchi
  - NISHIKAWA Women's Health Clinic, Sapporo

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/